CLINICAL TRIAL: NCT06612437
Title: Optimization of Time Parameters of Priming iTBS for Poststroke Motor Rehabilitation
Acronym: TMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Kenneth N. K. Fong, Prof., The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20240229006
Record Dates: First submitted 2024-09-21; First posted 2024-09-25 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Stroke Rehabilitation
Keywords: Stroke; TMS; TBS; EEG
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- cTBS primed iTBS with 3-minute interval (Experimental): short interval(3min) between cTBS and iTBS
  Interventions: Device: continuous theta burst stimulation (cTBS); Device: intermittent theta burst stimulation (iTBS); Device: Robot-assisted training
- cTBS primed iTBS with 10-minute interval (Experimental): experimental interval(10min) between cTBS and iTBS
  Interventions: Device: continuous theta burst stimulation (cTBS); Device: intermittent theta burst stimulation (iTBS); Device: Robot-assisted training
- cTBS primed iTBS with 20-minute interval (Experimental): long interval(20min) between cTBS and iTBS
  Interventions: Device: continuous theta burst stimulation (cTBS); Device: intermittent theta burst stimulation (iTBS); Device: Robot-assisted training
- Non-primed iTBS (Sham Comparator): iTBS alone
  Interventions: Device: intermittent theta burst stimulation (iTBS); Device: Robot-assisted training

INTERVENTIONS:
Device: continuous theta burst stimulation (cTBS) — Standard 600-pulse continuous theta burst stimulation (cTBS) can inhibit the corticomotor excitability. The cTBS will be delivered with an intensity of 70% individual resting motor threshold (RMT) of the hand knob over the contralesional M1.
  Other Names: Repetitive transcranial magnetic stimulation (rTMS)
  Arms: cTBS primed iTBS with 10-minute interval; cTBS primed iTBS with 20-minute interval; cTBS primed iTBS with 3-minute interval
Device: intermittent theta burst stimulation (iTBS) — Standard 600-pulse intermittent theta burst stimulation (iTBS) can increase the corticomotor excitability. The iTBS will be delivered with an intensity of 70% individual resting motor threshold (RMT) of the hand knob over the contralesional M1.
Device: Robot-assisted training — Fourier M2 upper limb rehabilitation robot (Fourier Intelligence Co. Ltd., Shanghai, China), will be used for upper limb proximal joints training. Fourier M2 upper limb rehab robot is an end-effector robot-assisted device. The device targets (1) flexion and extension of shoulder joint, (2) flexion and extension of elbow, (3) internal and external rotation of shoulder joint, and (4) abduction and adduction of shoulder joint, supported by tailored interactive TV games in the device.

SUMMARY:
The goal of this clinical trial is to identify the effect of different time intervals between continuous theta burst stimulation (cTBS) and intermittent theta burst stimulation(iTBS), on top of a standard robot-assisted training (RAT) for sensorimotor rehabilitation in patients with chronic stroke. Using electroencephalography (EEG) to explore potential sensorimotor neuroplasticity underying stroke.

DETAILED DESCRIPTION:
Delivering Intermittent theta burst stimulation (iTBS) primed with continuous theta burst stimulation (cTBS) to the primary motor cortex (M1) may enhance the facilitatory effect of iTBS on the stimulated M1 through metaplasticity. Previous studies have verified the effectiveness of priming iTBS on improving motor rehabilitation in patients with stroke. However, the optimal time interval between cTBS and iTBS remains unknown. The aim of this clinical trial is to identify the effect of different time intervals between cTBS and iTBS, followed with a standard robot-assisted training (RAT) for sensorimotor rehabilitation in patients with chronic stroke. Using electroencephalography (EEG) to explore potential sensorimotor neuroplasticity. A three-arm randomized controlled trial (RCT) will be performed with an estimated total of 30 patients with chronic stroke. All participants will be randomly allocated to receive 10-session intervention of different TBS protocols (i.e., cTBS-3min interval-iTBS, cTBS-10min interval-iTBS and cTBS-20min interval-iTBS), delivered for 2-4 sessions per week, lasting for 3-4 weeks. All participants will receive a 20-minute standard RAT after each stimulation session. Primary outcome will be Fugl-Meyer Assessment-Upper Extremity scores (FMA-UE). Secondary outcomes will be Action Research Arm Test (ARAT), kinematic outcomes generated during RAT as well as EEG.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of hemorrhagic or ischemic stroke using computed tomography (CT) or magnetic resonance imaging (MRI).
2. the first-ever stroke with unilateral hemiplegia.
3. 18-75 years old.
4. chronic stroke ( ≥ 6 months).
5. residual hemiparetic upper limb functional level in the Functional Test for the Hemiplegic Upper Extremity (FTHUE-HK) ≥ 2.
6. can understand and read Chinese.
7. signed informed consent.

Exclusion Criteria:

1. diagnosis of any clinically significant or unstable medical disorder.
2. any contraindications to TMS based on the TMS safety guidelines (Rossi, Hallett, Rossini, & Pascual-Leone, 2011).
3. inability to follow treatment instructions due to severe cognitive (using the Hong Kong version of the Montreal Cognitive Assessment (MoCA-HK) < 22/30) and communication deficiency.
4. extreme spasticity over the hemiparetic upper limb (Modified Ashworth Score>2) or severe pain that hindered movement.
5. a history of neurological or psychiatric disease excluding stroke, or current use of psychoactive medication (sedatives, antipsychotics, antidepressants, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer assessment of upper extremity (FMA-UE) | Baseline (Day 1, prior to first treatment), Day 21 (immediately after 10th treatment) , 1 month after completion of treatment
  Fugl-Meyer Assessment of upper extremity (FMA-UE) scale is an index to assess the sensorimotor impairment in individuals who have had stroke. It contains motor assessment and sensory assessment. The motor parts includes 33 items assessing the movement, coordination and reflex actions of the shoulder, elbow, forearm and wrist, as well as the hand joints of the paretic arm. Each item consists of a three-point scale (0, 1 and 2), with a total maximum score of 66. The sensory component consists of 6 items assessing light touch and position of the shoulder, elbow, wrist, and thumb. Each item consists of a three-point scale (0, 1, and 2) with a total score of 12 points.

SECONDARY OUTCOMES:
Action Research Arm Test (ARAT) | Baseline (Day 1, prior to first treatment), Day 21 (immediately after 10th treatment) , 1 month after completion of treatment
  The ARAT is a clinical assessment for upper limb functional activities for patients with stroke, which mainly focuses on the proximal and distal upper limb function. It consists of four subscales: grasp, grip, pinch and gross movement. It has 19 movement tasks, each graded using a four-point scale (total scores range from 0 to 57) (McDonnell, 2008). The MCID of ARAT is 5.70 points (Van der Lee et al., 2001).

OTHER OUTCOMES:
Sensorimotor event-related desynchronization | Baseline (Day 1, prior to first treatment), Day 1 (immediately after first treatment), Day 21 (immediately after 10th treatment)
  Electroencephalographical assessment for cortical activation induced by movement and mirror visual feedback-based observation of movement
Sensory evoked potential | Baseline (Day 1, prior to first treatment), Day 1 (immediately after first treatment), Day 21 (immediately after 10th treatment)
  Electroencephalographical assessment for cortical activation induced by periphral magenetic stimulation over the bilateral forearm.

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - The Hong Kong Polytechnic University, Hong Kong, HK
  - The Hong Kong Polytechnic University, Hong Kong

IPD SHARING:
Plan to Share IPD: No
To protect the privacy of patients

REFERENCES:
- [Result] Zhang JJ, Bai Z, Fong KNK. Priming Intermittent Theta Burst Stimulation for Hemiparetic Upper Limb After Stroke: A Randomized Controlled Trial. Stroke. 2022 Jul;53(7):2171-2181. doi: 10.1161/STROKEAHA.121.037870. Epub 2022 Mar 23. PMID 35317611